CLINICAL TRIAL: NCT06746363
Title: The Effectiveness of High-flow Nasal Cannula After Extubation in Patients
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Lo Tzu Han, Principal Investigator, Chang Gung Memorial Hospital
Other Study IDs: 202200799B0
Record Dates: First submitted 2024-11-29; First posted 2024-12-24 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Post Extubation Respiratory Failure
Keywords: post extubation; HFNC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HFNC group: HFNC support post extubation
- oxygen therapy: oxygen therapy post extubation

SUMMARY:
Observe the current status of prolonged mechanical ventilation (PMV) patients using high-flow nasal cannula oxygen therapy (experimental group) or traditional oxygen therapy (control group) after extubation, and compare the differences in ventilator weaning rates between the two groups.

Record the ROX index (SpO2/FiO2/RR) at 2, 6, 12, and 24 hours after extubation in PMV patients and explore whether statistical methods can predict the weaning outcome within seven days.

Use statistical methods to analyze whether comorbidities in the PMV population affect ventilator weaning rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 20 years old and expected to undergo extubation.

Exclusion Criteria:

* Patients with tracheostomy who will use non-invasive or invasive ventilators immediately after extubation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sample Size: The sample size was calculated using the G Power statistical software with a chi-square test. Parameters used were effect size: 0.3, alpha: 0.05, and power: 0.8. Based on these conditions, the required sample size is estimated to be 88 participants.
  Experimental Group: Comprising 44 PMV (Prolonged Mechanical Ventilation) patients who, after extubation, are assessed by physicians to use high-flow nasal cannula oxygen therapy.
  Control Group: Comprising 44 PMV patients who, after extubation, are assessed by physicians to use traditional oxygen therapy.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
ROX index | From enrollment to preliminary data compilation, lasting a total of 4 months.
  The oxygen concentration used before and after oxygen therapy adjustment is recorded as percent, accompanied by clinical and physiological parameter the patient's oxygen saturation (SpO₂) and respiratory rate (breaths per minute). Additionally, multiple measurements of the ROX index are performed, combining saturation (SpO₂), FiO₂, and respiratory rate to calculate and report the ROX index (SpO₂ / FiO₂ / RR).
P/F ratio | From enrollment to preliminary data compilation, lasting a total of 4 months.
  Collect the arterial oxygen partial pressure (PaO₂, mmHg) from each patient's clinical arterial blood dialysis, and compare it with the oxygen concentration (%) being used at the time. The two values are then combined to calculate the P/F ratio (PaO₂, mmHg / FiO₂, decimal).

OTHER OUTCOMES:
Area Under Curve (AUC) | From enrollment to the end of treatment at 1.5 year
  he Area Under the Curve (AUC) quantifies the overall performance of a model. The AUC ranges from 0 to 1, where an AUC of 0.5 indicates no discriminative power (random guessing), and an AUC of 1.0 indicates perfect discrimination that distinguishes between positive and negative classes without error.
  A higher AUC value suggests better model performance in distinguishing between classes, making it a widely used measure for assessing predictive accuracy in clinical and research datasets.
Receiver Operating Characteristic (ROC) curve | From enrollment to the end of treatment at 1.5 year
  the Receiver Operating Characteristic (ROC) curve, the performance of two predictive models, Logistic Regression and Random Forest, in predicting HFNC (High-Flow Nasal Cannula) weaning success. The curve plots the True Positive Rate (Sensitivity) on the y-axis against the False Positive Rate (1 - Specificity) on the x-axis across various classification thresholds.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
this study is the result of collaborative efforts by co-researchers.

REFERENCES:
- [Result] Fernandez R, Subira C, Frutos-Vivar F, Rialp G, Laborda C, Masclans JR, Lesmes A, Panadero L, Hernandez G. High-flow nasal cannula to prevent postextubation respiratory failure in high-risk non-hypercapnic patients: a randomized multicenter trial. Ann Intensive Care. 2017 Dec;7(1):47. doi: 10.1186/s13613-017-0270-9. Epub 2017 May 2. PMID 28466461
- [Result] Lee YS, Chang SW, Sim JK, Kim S, Kim JH. An Integrated Model including the ROX Index to Predict the Success of High-Flow Nasal Cannula Use after Planned Extubation: A Retrospective Observational Cohort Study. J Clin Med. 2021 Aug 10;10(16):3513. doi: 10.3390/jcm10163513. PMID 34441809
- [Result] Rochwerg B, Granton D, Wang DX, Helviz Y, Einav S, Frat JP, Mekontso-Dessap A, Schreiber A, Azoulay E, Mercat A, Demoule A, Lemiale V, Pesenti A, Riviello ED, Mauri T, Mancebo J, Brochard L, Burns K. High flow nasal cannula compared with conventional oxygen therapy for acute hypoxemic respiratory failure: a systematic review and meta-analysis. Intensive Care Med. 2019 May;45(5):563-572. doi: 10.1007/s00134-019-05590-5. Epub 2019 Mar 19. PMID 30888444
- [Result] Roca O, Messika J, Caralt B, Garcia-de-Acilu M, Sztrymf B, Ricard JD, Masclans JR. Predicting success of high-flow nasal cannula in pneumonia patients with hypoxemic respiratory failure: The utility of the ROX index. J Crit Care. 2016 Oct;35:200-5. doi: 10.1016/j.jcrc.2016.05.022. Epub 2016 May 31. PMID 27481760